CLINICAL TRIAL: NCT02410096
Title: Examination of Bronchial Inflammation and Hyperresponsiveness After Oil Supplementation With Middle-chain and Polyunsaturated Fatty Acids in an Exercise-induced Asthma Provocation Model
Brief Title: Bronchial Inflammation and Hyperresponsiveness After Oil Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Consultant Pediatric Allergy and Pneumology, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KGU-360/14
Record Dates: First submitted 2015-03-18; First posted 2015-04-07 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Exercise-induced Asthma
Keywords: exercise-induced asthma; cold chamber; exercise challenge; cold air challenge; oil supplementation; middle-chain and Polyunsaturated Fatty Acids
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oil supplementation verum (Active Comparator): 30 patients aged 12-44 years with a diagnosis of exercise induced asthma undergo a methacholine challenge and a prick test. After randomization patients will receive in double blind approach ones daily 1190 mg of middle-chain and polyunsaturated fatty acids for four weeks. Before and after supplementation an exercise challenge in a cold chamber will be performed.
  Interventions: Other: Exercise challenge in a cold chamber; Other: Methacholine challenge; Dietary Supplement: Oil supplementation verum
- Oil supplementation placebo (Placebo Comparator): 30 patients aged 12-44 years with a diagnosis of exercise induced asthma undergo a methacholine challenge and a prick test. After randomization patients will receive in double blind approach placebo for four weeks. Before and after placebo treatment an exercise challenge in a cold chamber will be performed.
  Interventions: Other: Exercise challenge in a cold chamber; Other: Methacholine challenge; Dietary Supplement: Oil supplementation placebo

INTERVENTIONS:
Other: Exercise challenge in a cold chamber — Exercise challenge is defined as running on a treadmill for 6-8 minutes on submaximal work load in a cold chamber.
Other: Methacholine challenge — Nebulized metacholine administered at following doses: 0,01mg, 0,1mg, 0,4mg, 0,8mg und 1,6mg
Dietary Supplement: Oil supplementation verum — Patients and subjects will take double blind an oil supplementation with middle-chain and polyunsaturated fatty acids for four weeks
  Arms: Oil supplementation verum
Dietary Supplement: Oil supplementation placebo — Patients and subjects will take double blind sunflower oil for four weeks
  Arms: Oil supplementation placebo

SUMMARY:
The purpose of this study is to investigate the bronchial inflammation and hyperresponsiveness after oil supplementation. Before and after oil supplementation the investigators measure decrease in lung function after exercise-challenge in a cold chamber and increase of inflammatory markers in the blood.

DETAILED DESCRIPTION:
Subjects suffering form exercise-induced bronchoconstriction (EIB) usually have a normal lung function testing at rest and show a decrease in lung function when they do sports or an exercise-challenge. In a previous study the investigators could show, that the combination of exercise test and inhalation of cold air ist more sensitive and specific than exercise-challenge in ambient temperature.

It is known that omega - 3 -fatty acids could reduce the production of inflammatory mediators.

In this study the investigators will investigate the protective effect of oil supplementation with middle-chain and polyunsaturated fatty acids in an exercise-induced asthma provocation model.

Therefore the investigators will measure the decrease in lung function and a increase of inflammatory markers in the blood before and after oil supplementation.

Before and after the exercise-challenge the investigators will measure spirometry and body plethysmography. The investigators want to examine if the body plethysmography is more sensitive in the measurement of exercise induced bronchoconstriction than spirometry.

The investigators hypothesize that the oil supplementation can reduce bronchial inflammation and hyperresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients: Age ≥12 and 44 years
* known exercise induced asthma
* basic lung function FVC ≥ 75%, FEV1 ≥ 70%
* decrease in FEV1 after exercise ≥ 15%

Exclusion Criteria:

* lung function Forced vital capacity (FVC) <75% and Forced expiratory volume in 1 second (FEV1) <70%
* chronic diseases or infections (e.g. HIV, Tbc)
* pregnancy
* systemic corticosteroid-treatment
* inhalative corticosteroid therapy or leukotriene antagonists
* alcohol, substance or drug abuse
* smokers
* inability to capture extend and consequences of the study

Ages: 12 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Decrease in FEV1 after exercise challenge in cold air as measured by spirometry (FEV1, percent predicted) - comparison verum vs placebo | 4 weeks
  The exercise challenge in cold air will be done on two timepoints. Before and after oil supplementation versus placebo supplementation. After exercise challenge spirometry will be measured. Decrease in FEV1 in verum and control group will be compared with t-test and Wilcoxon-Mann-Whitney-Test.

SECONDARY OUTCOMES:
Comparison of decrease in exhaled nitric oxide (eNO) as measured by Niox Mino (parts per billion, ppb) | 4 weeks
  Comparison of decrease in eNO before and after supplementation in verum and placebo group
Comparison of change in lipids in serum as measured by capillary gas chromatography (weight percent, wt%) | 4 weeks
  Comparison of increase eicosapentaenoic acid and docosahexaenoic acid and decrease of triglycerides before and after supplementation in verum and placebo group

OTHER OUTCOMES:
Comparison of two methods of lung function testing as measured by spirometry (FEV1, percent predicted) and body plethysmography (specific airway resistance, sRAW, kPa*sec) | 4 weeks
  Both methods will be done in parallel before and 4 times after exercise challenge in cold air. Afterwards the investigators can compare both methods and calculate the sensitivity for both methods to indicate exercise induced bronchoconstriction.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schulze, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Schubert R, Kitz R, Beermann C, Rose MA, Lieb A, Sommerer PC, Moskovits J, Alberternst H, Bohles HJ, Schulze J, Zielen S. Effect of n-3 polyunsaturated fatty acids in asthma after low-dose allergen challenge. Int Arch Allergy Immunol. 2009;148(4):321-9. doi: 10.1159/000170386. Epub 2008 Nov 11. PMID 19001792
- [Background] Schulze J, Smith HJ, Fuchs J, Herrmann E, Dressler M, Rose MA, Zielen S. Methacholine challenge in young children as evaluated by spirometry and impulse oscillometry. Respir Med. 2012 May;106(5):627-34. doi: 10.1016/j.rmed.2012.01.007. Epub 2012 Feb 10. PMID 22326606
- [Background] Nensa F, Kotschy-Lang N, Smith HJ, Marek W, Merget R. Assessment of airway hyperresponsiveness: comparison of spirometry and body plethysmography. Adv Exp Med Biol. 2013;755:1-9. doi: 10.1007/978-94-007-4546-9_1. PMID 22826043
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563
- [Background] Dyerberg J, Bang HO. Lipid metabolism, atherogenesis, and haemostasis in Eskimos: the role of the prostaglandin-3 family. Haemostasis. 1979;8(3-5):227-33. doi: 10.1159/000214314. PMID 511010
- [Background] Endres S, Ghorbani R, Kelley VE, Georgilis K, Lonnemann G, van der Meer JW, Cannon JG, Rogers TS, Klempner MS, Weber PC, et al. The effect of dietary supplementation with n-3 polyunsaturated fatty acids on the synthesis of interleukin-1 and tumor necrosis factor by mononuclear cells. N Engl J Med. 1989 Feb 2;320(5):265-71. doi: 10.1056/NEJM198902023200501. PMID 2783477
- [Background] Mickleborough TD, Murray RL, Ionescu AA, Lindley MR. Fish oil supplementation reduces severity of exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Nov 15;168(10):1181-9. doi: 10.1164/rccm.200303-373OC. Epub 2003 Aug 6. PMID 12904324
- [Background] Parsons JP, Hallstrand TS, Mastronarde JG, Kaminsky DA, Rundell KW, Hull JH, Storms WW, Weiler JM, Cheek FM, Wilson KC, Anderson SD; American Thoracic Society Subcommittee on Exercise-induced Bronchoconstriction. An official American Thoracic Society clinical practice guideline: exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2013 May 1;187(9):1016-27. doi: 10.1164/rccm.201303-0437ST. PMID 23634861
- [Derived] Dressler M, Fussbroich D, Bohler L, Herrmann E, Benker N, Tytyk M, Schulze J, Schubert R, Beermann C, Zielen S. Oil supplementation with a special combination of n-3 and n-6 long-chain polyunsaturated fatty acids does not protect for exercise induced asthma: a double-blind placebo-controlled trial. Lipids Health Dis. 2020 Jul 13;19(1):167. doi: 10.1186/s12944-020-01343-2. PMID 32660564